CLINICAL TRIAL: NCT01358994
Title: Metformin Treatment, Renal Function and Lactic Acidosis. A Population Based
Brief Title: Metformin Treatment, Renal Function and Lactic Acidosis
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Gunnar Sterner, PhD, Skane University Hospital
Other Study IDs: Metformin02
Record Dates: First submitted 2011-05-19; First posted 2011-05-24 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: metformin; type 2 diabetes; e-GFR; creatinine; lactic acidosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Acidosis, Lactic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
From a central registry at the National Board of Health and Welfare in Sweden collect all patients in the city of Malmö prescribed metformin during two years. Glomerular filtration rate (eGFR) was estimated from the CKD-EPI formula (n=5408) and compared to a control material (n=2815) from the same town. All cases of severe lactic acidosis rendering ICU admission were also sought. The study hypothesis is that metformin is prescribed to patients with lower GFR than anticipated with very few cases of lactic acidosis registered.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the city of Malmö prescribed metformin at least three times during two years
* Available at least one p-creatinine during the two years

Exclusion Criteria:

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients irrespective of age prescribed metformin according to a registry for the city of Malmö
Sampling Method: Probability Sample
Enrollment: 4500 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Nephrology, Malmo, Sweden